CLINICAL TRIAL: NCT03243149
Title: Neurofeedback With Real-Time fMRI for Treatment of Posttraumatic Stress Disorder
Brief Title: Neurofeedback With Real-Time fMRI for Treatment of PTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient staff and equipment challenges
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00081664
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The investigators will test (1) the efficacy of neurofeedback in subjects with PTSD attempting to upregulate ventral medial PFC and simultaneously downregulate amygdala, and (2) determine the number of neurofeedback sessions (dose) needed for target engagement and transfer. Prior to the neurofeedback training, participants' baseline ability to regulate in the absence of neurofeedback from real-time fMRI will be ascertained. Then during session, participants will receive veridical real-time feedback in the scanner indicating the activation level of ventromedial PFC minus amygdala. Participants will attempt to regulate to achieve a predetermined target level known to the participant.
Who Masked: Participant
Masking Description: Participants will be unaware of whether the thermometer ratings they see while in the scanner are false feedback consisting of noise or true activation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- False Feedback (Sham Comparator): Neurofeedback from real-time acquired images (fMRI - GE Medical System) will be shown to subjects. False feedback (sham) shows a thermometer that indicates false feedback consisting of noise.
  Interventions: Device: fMRI - GE Medical System
- View Condition (Active Comparator): Neurofeedback from real-time acquired images (fMRI - GE Medical System) will be shown to subjects. View condition shows a thermometer that indicates true activation of ventromedial PFC minus amygdala but the participant is asked not to attempt neuroregulation.
  Interventions: Device: fMRI - GE Medical System
- Free Regulate (Experimental): Neurofeedback from real-time acquired images (fMRI - GE Medical System) will be shown to subjects. Free regulate shows a thermometer that indicates true activation of ventromedial PFC minus amygdala while the participant attempts neuroregulation.
  Interventions: Device: fMRI - GE Medical System

INTERVENTIONS:
Device: fMRI - GE Medical System — Recovery from PTSD symptoms has been modeled experimentally as fear extinction that depends on three interconnected brain regions that involve the amygdala where extinction memories are stored, the subcallosal/subgenual cortex within the medial PFC involved in consolidation of the extinction memory, and the hippocampus which mediates the context specificity of context specificity of extinction.
  The two MRI systems are used for human research by many faculty and research groups at Duke and UNC, Chapel Hill. The center has two research dedicated General Electric MR 750 scanners with a field strength of 3 Tesla. These systems use a combination of General Electric production pulse sequences and custom research pulse sequences that have been developed by Brain Imaging and Analysis Center faculty and other MR physicists. The scanners are used for imaging and spectroscopy.
  Other Names: Neurofeedback regulation of fear extinction neurocircuitry

SUMMARY:
PTSD is a debilitating and costly condition and currently available treatment options have risks and limitations that necessitate development of novel interventions. Collectively, the functional brain imaging reports suggest that patients with PTSD, especially those with the re-experiencing and hypervigilence phenotype, show ventromedial PFC hypoactivation and amygdala hyperactivation in response to symptom provocation, and that treatment, when successful is associated with reduced amygdala and increased ventromedial PFC activation. This project is guided by a neurocircuit model of PTSD dysfunction in which abnormalities in fronto-limbic imbalance, which diminishes capacity for fear extinction learning, and produces PTSD symptoms of re-experiencing and hyperarousal. Thus, our studies aim to bridge the translational gap between theoretical and neurobiological models of PTSD to implementation of clinical practice. The Target Engagement and Dosing Phase of this project, which is a pilot study, will demonstrate target engagement and its association with laboratory measures of PTSD-relevant neural processes.

DETAILED DESCRIPTION:
The proposed treatment is expected to reduce symptoms of PTSD particularly re-experiencing and hyperarousal symptoms. These improvements in symptoms are expected to translate into improved social and occupational function for subjects with PTSD.

Specific Aim 1: The investigators will test (1) the efficacy of neurofeedback in subjects with PTSD attempting to upregulate ventral medial PFC and simultaneously downregulate amygdala, and (2) determine the number of neurofeedback sessions (dose) needed for target engagement and transfer. Prior to the neurofeedback training, participants' baseline ability to regulate in the absence of neurofeedback from real-time fMRI will be ascertained. Then during session, participants will receive veridical real-time feedback in the scanner indicating the activation level of ventromedial PFC minus amygdala. Participants will attempt to regulate to achieve a predetermined target level known to the participant. Neurofeedback conditions will include (1) false feedback (sham) shows a thermometer that indicates false feedback consisting of noise, (2) view condition shows a thermometer that indicates true activation of ventromedial PFC minus amygdala but the participant is asked not to attempt neuroregulation, (3) free regulate shows a thermometer that indicates true activation of ventromedial PFC minus amygdala while the participant attempts neuroregulation. The investigators will enroll 10 participants who will engage in a six weekly neurofeedback sessions to assess target engagement and dosing.

Specific Aim 2: The ability for participants to regulate will be further challenged by explicit exposure to trauma relevant stimuli that elicit increased amygdala activation in patients with PTSD. The investigators will follow the same procedure as the previous aim except that free regulate condition (condition #3) will be replaced with conditions (4) trauma regulate shows a participant-specific trauma-relevant image and the thermometer that indicates true activation of ventromedial PFC minus amygdala while the participant attempts neuroregulation, and (5) neutral regulate shows a trauma-unrelated image and the thermometer that indicates true activation of ventromedial PFC minus amygdala while the participant attempts neuroregulation. The investigators will enroll 10 participants who will engage in a six weekly neurofeedback sessions to assess target engagement and dosing.

Participants will be assessed for PTSD and related symptoms before and after to the 6-week intervention using the Clinician Administered PTSD Scale (CAPS) (Appendix XVI) and Beck Depression Inventory (BDI-II) (Appendix IX). The investigators hypothesize enhanced neuroregulation and transfer will be associated with a concomitant reduction in PTSD severity and lower comorbid anxiety symptoms.

Specific Aim 3: Participants will be assessed before and after the 6-week intervention with a brief neurocognitive battery of episodic memory, working memory, executive function, and sustained attention. The investigators hypothesize that successful neuroregulation and transfer will be associated with concomitant cognitive performance improvements.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English and capable of informed consent
* free of implanted metal objects
* 18-50 years of age
* Antidepressant sleep and anti-anxiety medication use is permitted

Exclusion Criteria:

* Claustrophobia
* Neurological disorders, History of learning disability or developmental delay
* Current substance abuse or history of substance dependence
* Psychotic disorders
* Significant medical conditions
* Current suicidality or attempt within the previous year
* History of neurological injury or disease
* Pregnancy
* Major Axis 1 Psychiatric Disorders (exceptions are unipolar depression, past substance abuse, current or past nicotine dependence)
* Metal in the body

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Change in MRI Imaging Acquisition | Baseline scan (week 1), week 2, week 3, week 4, week 5 and week 6.
  fMRI scans will use a 3T GE scanner at the Duke-UNC Brain Imaging and Analysis Center. Structural MRI data and functional MRI data that includes real-time feedback on the participants brain activity will be made available to the participant to facilitate self-regulation.
  Participants will begin and end each scanning session with a 6-minute resting-state scan. The purpose of the first resting-state run is collect pre-Training baseline resting-state activation and to acclimate the subject to the scanner environment prior to neuroregulatory training. The purpose of the second resting state run is examine changes in functional connectivity after compared to before real-time fMRI neurofeedback.
  To determine the effect of session on subject ability to increases ventromedial prefrontal cortex activation and decrease amygdala activation and establish a dose-response relationship for neuroregulation, we will measure changes in BOLD signal across scan sessions.

SECONDARY OUTCOMES:
Change in psychophysiological data | Baseline scan (week 1), week 2, week 3, week 4, week 5 and week 6.
  Physiological measures of heart rate and respiration will be recorded during each scan, using an MR-safe commercial system (MP-150 BIOPAC systems, Goleta, CA) to permit removal of physiological noise from the fMRI signal. To evaluate potential scalable non-fMRI correlates, we will also acquire pupillometry using an MR-compatible camera (Arrington Research, Inc.) and galvanic skin conductance levels to identify fear or anxiety responses that impede self-activation.
  To determine the effect of session on subject ability to regulate stress through neurofeedback, we will measure changes in psychophysiological data across scan sessions.
Change in Clinician Administered PTSD Scale (CAPS) Severity Score | Baseline, 6 weeks
  Participants will be assessed for current and lifetime PTSD twice, once at the beginning and once at the end of the 6 weeks.
Beck Depression Inventory-II (BDI-II) | Baseline
  Diagnostic assessment for PTSD and comorbid symptoms of depression
Drug Abuse Screening Test (DAST) | Baseline
  Diagnostic assessment for substance use
Combat Exposure Scale (CES) | Baseline
  Diagnostic assessment for combat exposure.
Deployment Risk and Resilience Inventory-2 (DRRI-2) | Baseline
  Baseline diagnostic assessment for both risk and resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra A Morey, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
Except when required by law, the investigators will not identify subjects by name, social security number, address, telephone number, or any other personal identifier in study records disclosed outside DUMC. For records disclosed outside DUMC, only the subjects' identification numbers will be used. Coded data that includes MRI images, MRI task based responses, psychometric, and diagnostic information will be released to collaborating investigators. The study results will be retained in subjects' research records for an indefinite time after completion of the study.